CLINICAL TRIAL: NCT02996227
Title: Comparison of Bilateral Transversus Abdominis Plane Block With Exparel Verus Continuous Epidural Analgesia With Bupivacaine: A Randomized, Controlled Trial
Brief Title: Bilateral Transversus Abdominis Plane Block With Exparel Verus Continuous Epidural Analgesia With Bupivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1449 -EXPLANE Block
Record Dates: First submitted 2016-12-05; First posted 2016-12-19 (Estimated); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Pain, Postoperative; Major Abdominal Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Epidural; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP block with Exparel (Experimental): Bilateral Transversus Abdominis Plane (TAP) block procedure following injection of liposomal bupivacaine (Exparel)
  Interventions: Procedure: TAP block; Drug: EXPAREL
- Epidural analgesia with Bupivacaine (Active Comparator): Epidural catheters with an infusion of Bupivacaine standard solution without additives
  Interventions: Procedure: Epidural analgesia; Drug: Bupivacaine

INTERVENTIONS:
Procedure: TAP block — Transversus Abdominis Plane (TAP) blocks will be performed preoperatively. An in-plane ultrasound will be used in TAP block procedure.
  Arms: TAP block with Exparel
Procedure: Epidural analgesia — Epidural catheters will be inserted preoperatively.
  Arms: Epidural analgesia with Bupivacaine
Drug: EXPAREL — Once the target area is positioned, plain bupivacaine 0.25%, 20ml will be given to open the space and then single dose (10ml) of liposomal bupivacaine (Exparel) mixed with saline (10 ml) will be injected in each side. Total dose of Exparel will be 20 mL.
  Other Names: Liposomal Bupivacaine
  Arms: TAP block with Exparel
Drug: Bupivacaine — Once an epidural catheter is successfully positioned, an infusion will be initiated intraoperatively. Bupivacaine standard solution without additives will be prepared for each patient in epidural group.
  Other Names: Marcaine
  Arms: Epidural analgesia with Bupivacaine

SUMMARY:
Comparison of Bilateral Transversus Abdominis Plane Block with Exparel versus Continuous Epidural Analgesia With Bupivacaine

DETAILED DESCRIPTION:
The investigator goal is to compare the analgesic efficacy of TAP blocks with liposomal bupivacaine (Exparel) and continuous epidural blocks in patients who are scheduled for major lower abdominal surgery. To assess whether TAP block with Exparel is noninferior to continuous epidural analgesia on pain management, defined as noninferior for both pain control and total opioid consumption for 72 hours, in patients who had major lower abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* 18-85 years old
* ASA Physical Status 1-3
* Scheduled for elective open or laparoscopic abdominal surgery, including colorectal and hysterectomy surgeries
* Anticipated hospitalization of three nights
* Expected requirement for parenteral opioids for at least 72 hours for postoperative pain
* Able to use IV PCA systems.

Exclusion Criteria:

* Hepatic disease, e.g. twice the normal levels of liver enzymes
* Kidney disease, e.g. twice the normal level of serum creatinine
* Bupivacaine sensitivity or known allergy
* Women who are pregnant or breastfeeding
* Anticoagulants considered to be a contraindication for epidural or TAP blocks.
* Surgeries with high port sites will be excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2016-12; Primary Completion 2019-06 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Derived] Turan A, Cohen B, Elsharkawy H, Maheshwari K, Soliman LM, Babazade R, Ayad S, Hassan M, Elkassabany N, Essber HA, Kessler H, Mao G, Esa WAS, Sessler DI; EXPLANE Study Group. Transversus abdominis plane block with liposomal bupivacaine versus continuous epidural analgesia for major abdominal surgery: The EXPLANE randomized trial. J Clin Anesth. 2022 May;77:110640. doi: 10.1016/j.jclinane.2021.110640. Epub 2021 Dec 27. PMID 34969004

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
Started | 260 | 254
Completed | 255 | 243
Not Completed | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine | Total
Number analyzed (Participants) | 255 | 243 | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14) | 56 (14) | 55 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 161 | 321
  Male | 95 | 82 | 177
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 221 | 213 | 434
  Other | 34 | 30 | 64
ASA Status [Count of Participants; unit: Participants] — Patients were categorized among the 4 ASA physical status according to the pre-anesthesia appointment. This classification uses a grading system of I (better) until IV (worse).
  ASA I: A normal healthy patient ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life.
  Participants
    I | 2 | 2 | 4
    II | 70 | 67 | 137
    III | 171 | 167 | 338
    IV | 12 | 6 | 18
    Unknown | 0 | 1 | 1
Procedure type [Count of Participants; unit: Participants]
  Open | 188 | 181 | 369
  Laparoscopic | 67 | 62 | 129
Surgery Duration [Mean (Standard Deviation); unit: hours] | 5.7 (2.5) | 5.6 (2.5) | 5.7 (2.5)
Type of Surgery [Count of Participants; unit: Participants]
  Bariatric | 0 | 1 | 1
  Colorectal | 171 | 167 | 338
  Gynecologica | 55 | 42 | 97
  Urological | 2 | 5 | 7
  Other | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: VRS Pain Score
Description: Pain scores will be measured using a Verbal Response Scale (VRS). VRS is a scale from 0 to 10 where 0 signifies no pain and 10 signifies the worst pain ever experienced. The VRS will be recorded every 4 hours for 72 hours after discharge from the PACU. Summary statistics of pain scores are reported as means ± standard deviations of average pain during the first 72 postoperative hours
Time Frame: The Verbal Response Scale was recorded every 4 hours for 72 hours after discharge from the PACU.
Population: Two patients had missing outcomes due to the cancellation of surgery in Epidural analgesia with Bupivacaine group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
Number analyzed (Participants) | 255 | 241
score on a scale | 4.3 (1.8) | 4.2 (1.8)
Statistical Analysis 1: Comparison: TAP Block With Exparel vs Epidural Analgesia With Bupivacaine; Test type: Non-Inferiority — The noninferiority was defined as no more than 25% greater opioid consumption and no worse than 1-point higher pain score at rest. Non-inferiority of TAP with liposomal bupivacaine to epidural could be claimed if the upper limit of the 95.2% CI for the mean difference of pain scores at rest was less than 1 point and the CI for the ratio of geometric means in opioid consumption was less than 1.25; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95.2% CI 2-sided [-0.12 to 0.30]

2. Primary Outcome: Total Opioid Consumption
Description: Opioid consumption will be measured as the total amount of opioids (converted to morphine sulfate equivalents) used during the 72 hours after the end of surgery.
Time Frame: During the 72 hours after discharge from the PACU.
Population: Two patients had missing outcomes due to the cancellation of surgery in Epidural analgesia with Bupivacaine group.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
Number analyzed (Participants) | 255 | 241
mg | 56 [20 to 122] | 35 [13 to 94]
Statistical Analysis 1: Comparison: TAP Block With Exparel vs Epidural Analgesia With Bupivacaine; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.754, Mixed Models Analysis; Ratio of Geometric means = 1.37, 95.2% CI 2-sided [1.05 to 1.79]

3. Secondary Outcome: Cumulative Duration of Activity
Description: defined as the total duration of time patients spent sitting or standing, as determined by the mobile monitoring system during the initial 72 postoperative hours.
Time Frame: During the initial 72 postoperative hours.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
Number analyzed (Participants) | 123 | 118
hours | 1.1 [0.2 to 3.4] | 1.0 [0.1 to 3.8]
Statistical Analysis 1: Comparison: TAP Block With Exparel vs Epidural Analgesia With Bupivacaine; Test type: Superiority; p = 0.560, Regression, Linear; linear regression after logarithm transformation; Mean Difference (Final Values) = 1.2, 99% CI 2-sided [0.53 to 2.76]

4. Secondary Outcome: Opioid-related Side Effect
Description: We will use 4-point Opioid-Related Symptom Distress Scale (ORSDS) to evaluate the frequency, severity, and bothersomeness of: nausea, vomiting, constipation, difficulty passing urine, difficulty concentrating,drowsiness or difficulty staying awake, feeling lightheaded or dizzy,feeling confused, feelings of general fatigue or weakness, itchiness, dry mouth, and headache. Severity: 1=Slightly severe 2=Moderately severe 3=Severe 4=Very severe; Frequency: 1=Rarely 2=Occasionally 3=Frequently 4=Almost constantly; Bothersomeness (rescaled to a 4-point scale): 0.8=not at all 1.6=a little bit 2.4= somewhat 3.2=quite a bit 4.0=very much. If a patient did not experience the symptom in the past 24 hours, a score of 0 was assigned to each domain. Opioid-related side effect is the sum of the patient's frequency, severity, and bothersomeness, scored from 0 to 12. Higher scores indicate greater severity.
Time Frame: The first, second and third postoperative mornings
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
Number analyzed (Participants) | 203 | 199
score on a scale
  POD 1 | 5.8 [2.3 to 9.7] | 5.5 [2.8 to 9.6]
  POD 2 | 4.9 [1.9 to 9.1] | 4.5 [1.3 to 8.4]
  POD 3 | 3.8 [1.5 to 8.3] | 3.7 [0.9 to 8.7]
Statistical Analysis 1: Comparison: TAP Block With Exparel vs Epidural Analgesia With Bupivacaine; Test type: Superiority; p = 0.357, Regression, Linear; Mean Difference (Final Values) = 0.36, 99% CI 2-sided [-0.65 to 1.37] — Difference in means between two groups was assessed using mixed effects model with repeated measurements with unstructured correlation structure

5. Secondary Outcome: Hemodynamic Instability, Defined as Mean Arterial Pressure (MAP) <55 mmHg or Systolic Blood Pressure <80 mmHg.
Description: Visi mobile patient monitoring system will be used to obtain the blood pressure of the patient for 72 hours. Data was recorded at 15-s intervals and downloaded daily to a laptop. We re-defined postoperative hypotension as any MAP <65 mmHg, because few patients experienced such profound hypotension as originally planned and because papers published since the trial were designed to identify 65 mmHg as the harm threshold for both myocardial and renal injury. Summary statistics of hemodynamic instability are reported as means ± standard deviations of average MAP during the first 72 postoperative hours.
Time Frame: Data was recorded at 15-s intervals during the initial 72 postoperative hours.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
Number analyzed (Participants) | 123 | 119
mmHg | 41 (31) | 57 (48)
Statistical Analysis 1: Comparison: TAP Block With Exparel vs Epidural Analgesia With Bupivacaine; Test type: Superiority; p = 0.006, generalized linear regression; Risk Ratio (RR) = 0.64, 99% CI 2-sided [0.42 to 0.98]

6. Secondary Outcome: Quality of Recovery After Anesthesia
Description: Quality of recovery (QoR) will be measured using QoR-15 questionnaire which includes 15 11-point numerical rating scale. For positive items, 0 = "none of the time [poor]" to 10 = "all of the time [excellent]"; Conversely, for negative items, 10 = "none of the time [excellent]" to 0 = "all of the time [poor]". Quality of recovery is the sum of all the 15 questions, with a score ranging from 0 (extremely poor QoR) to 150 (excellent QoR).
Time Frame: The first and third postoperative mornings
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
Number analyzed (Participants) | 203 | 198
score on a scale
  POD 1 | 102 (26) | 100 (24)
  POD 3 | 111 (23) | 111 (22)
Statistical Analysis 1: Comparison: TAP Block With Exparel vs Epidural Analgesia With Bupivacaine; Test type: Superiority; p = 0.695, Regression, Linear; Mean Difference (Final Values) = 0.77, 99% CI 2-sided [-4.31 to 5.85] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Length of Hospital Stay
Description: The length of hospital stay will be measured as days.
Time Frame: From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 100 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
Number analyzed (Participants) | 255 | 241
days | 4.0 [3.0 to 7.0] | 4.0 [3.0 to 7.0]
Statistical Analysis 1: Comparison: TAP Block With Exparel vs Epidural Analgesia With Bupivacaine; Test type: Superiority; p = 0.738, Regression, Linear; linear regression after logarithmic transformation; Ratio of geometric means = 0.98, 99% CI 2-sided [0.86 to 1.12]

8. Other Pre Specified Outcome: Duration of Hypoxemia
Description: ViSi mobile (Sotera Wireless) patient monitoring system will be used to obtain vital signs including SpO2 of the patient for 72 hours. Data was recorded at 15-s intervals and downloaded daily to a laptop. The outcome is area-under-the-curve for saturation over time with the threshold set at 90%.
Time Frame: Data was recorded at 15-s intervals during the initial 72 postoperative hours.
Measure: Median (Inter-Quartile Range); unit: min/h
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
Number analyzed (Participants) | 123 | 118
min/h | 1.4 [0.2 to 7.7] | 2.8 [0.3 to 8.4]

9. Other Pre Specified Outcome: Persistent Postoperative Incisional Pain- MBPI Pain Intensity
Description: Defined by the presence of pain at three months and its characteristics as determined by Modified Brief Pain Inventory (MBPI) questionnaires. The modified BPI contains 4 intensity items and 5 interference items with 0-to-10 numerical rating scales. For intensity items: 0 = "no pain" and 10 = "pain as bad as you can imagine."; and for interference items, 0 = "does not interfere" and 10 = "interferes completely." The pain intensity is the sum of the patient's worst, average, least, and current pain intensity, with a score ranging from 0 (no pain) to 40 (pain as bad as you can imagine); and pain Interference is the sum of walking ability, mood, sleep, relations with others, and ability to concentrate, with a score ranging from 0 (does not interfere) to 50 (interferes completely).
Time Frame: At the 90-day follow up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
Number analyzed (Participants) | 59 | 54
score on a scale | 8 [5 to 17] | 12 [5 to 21]

10. Other Pre Specified Outcome: Persistent Postoperative Incisional Pain- MBPI Pain Interference
Description: as for outcome 9
Time Frame: At the 90-day follow up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
Number analyzed (Participants) | 59 | 54
score on a scale | 14 [3 to 34] | 17 [0 to 38]

ADVERSE EVENTS:
Time Frame: During the initial postoperative 3 months
Arm/Group | TAP Block With Exparel | Epidural Analgesia With Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/255 | 0/243
Serious Adverse Events (participants affected / at risk) | 0/255 | 0/243
Other Adverse Events (participants affected / at risk) | 0/255 | 0/243

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT02996227/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT02996227/ICF_001.pdf